CLINICAL TRIAL: NCT05267756
Title: Exploring the Difference in Using Virtual Reality Fully Immersive Based Exercise Game or Usual Care on Physical and Psychosocial Factors in People With Chronic Non-specific Low Back Pain
Brief Title: Effect Virtual Reality Fully Immersive Based Exercise Game on Reducing Fear of Movement in People With CLBP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, kholoud abdullah Almufaireej, Therapist, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VR with LBP
Record Dates: First submitted 2022-02-24; First posted 2022-03-04 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: CLBP - Chronic Low Back Pain
Keywords: CLBP; VR; Fear of movement; Disability; Video Game; Adherence
MeSH Terms: conditions — Kinesiophobia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention Group (Experimental): Patient will be receive .
  1. usual care that included the education patients(e.g., information, and behavior modification advice techniques) based on the latest clinical practice guidelines (Qaseem et al., 2017 ; Delitto et al., 2012). Also, Patients understood their back problem by reassurance that the condition is not a serious disease and information about the nature of the disorder and prognosis and course of recovery. And what should be done to reduce worry (e.g., stay active and returning to normal activities as soon as possible, avoid worry, coping with having a sore back, and positive attitudes towards back pain are important). The given pamphlets produced by the Saudi Spine Society.
  2. The intervention group will have in addition to the usual care, virtual reality immersive based-exercise game, the participants will download (kurki-application), and will given VR glasses
  Interventions: Device: (kurki-application),VR glasses
- Control Group (No Intervention): Patient will be receive .
  1. usual care that included the education patients(e.g., information, and behavior modification advice techniques) based on the latest clinical practice guidelines (Qaseem et al., 2017 ; Delitto et al., 2012). Also, Patients understood their back problem by reassurance that the condition is not a serious disease and information about the nature of the disorder and prognosis and course of recovery. And what should be done to reduce worry (e.g., stay active and returning to normal activities as soon as possible, avoid worry, coping with having a sore back, and positive attitudes towards back pain are important). The given pamphlets produced by the Saudi Spine Society.
  2. The control group will have in addition to usual care that included the education patients, a Brochure for LBP therapeutic exercises

INTERVENTIONS:
Device: (kurki-application),VR glasses — it is virtual reality immersive based-exercise game
  Arms: intervention Group

SUMMARY:
Low back pain is one of the most common problems among adults and a leading cause of disability worldwide including in Saudi Arabia (Buchbinder et al., 2018) (Awaji, 2016) . Studies have shown that 80% of adults would experience low back pain at least once in their lifetime (Awaji, 2016). Research has shown that physical exercises are the most effective rehabilitation method. However, some CLBP patients have fear of movement and fear of increasing the pain (Alamam et al., 2019b), which will lead to inactivity and more disability. Moreover, low adherence to the prescribed exercise program is very common, which could be due to complexity of the program, boredom or lack of supervision and follow up(Elbur, 2015). VR fully-immersive -based exercise game can be used to enhance CLBP rehabilitation by keeping the patients engaged in the virtual environment distracting them from pain and stopping the cycle of fear of movement. Based on the previous problem our research questions are:

* Will the VR fully immersive based exercise game improve patient outcomes (fear, pain, reduce disability and improves physical function and adherence)? Aims of the Study.
* To assess the effectiveness of the VR fully immersive-based exercise game in the rehabilitation program for patients with CNSLBP with kinesiophobia, in reducing fear of movement, pain-related to disability, and improving physical function.

To assess the adherence of the VR-based exercise, which has entertainment aspect is better than adherence to the conventional paper-based exercise.

DETAILED DESCRIPTION:
Significance of the Study. Based on the Fear-Avoidance model, the fear comes from the pain perception which increases level of disability (Leeuw et al., 2007). Thus, to break the fear cycle, we need first to reduce the pain intensity. This can be done by a virtual environment into a Head Mounted Displays (HMDs) that provides a fully immersive experience to engage the patients in a virtual environment and distract them from the pain while performing their exercises. Moreover, based on recent clinical guidelines for LBP rehabilitation, exercises are one of the most effective treatments for LBP. Therefore, we believe that a fully immersive based exercise game integrated with physical exercises that include a series of trunk movements such as moving forward, backward, sideways, and rotation. This solution will enhance the rehabilitation outcome since the patients who are suffering from CLBP with fear of movement and high level of disability can use the system at their home and train more for long period of time using a low-cost virtual reality device.

ELIGIBILITY:
Inclusion Criteria:

1. Consented adult patients, male and female, aged 18 or older.
2. patient diagnosed with chronic non-specific low back pain (symptoms duration more than 3 month).
3. patient reported no health condition that would restrict movement or prevent safe participation
4. patient able to use smart phone.

Exclusion Criteria:

1. patients age more than 60 years. (As patient has high risk of morbidity could affect balance and movement)
2. Patients with spine surgery, hip arthroplasty, or spinal deformity like scoliosis.
3. Patient with red flags (e.g., active cancer, report recent or unexplained loss weight, infection, inflammation, or fracture)
4. Clinical neurological features like lumbar radiculopathy.
5. vestibular system dysfunction like vertigo or imbalance by using Head impulse test(Furman & Barton, 2015).
6. pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-10-10 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Fear-avoidance Belief Questionnaire (FABQ) | The change after 2 weeks of intervention
  Consists of 16 items a self-report questionnaire based on evaluation on the Fear-avoidance model.The maximum score is 96, that representing higher levels of fear-avoidance beliefs. The FABQ has two subscales: the work subscale (FABQw),and the physical activity subscale (FABQpa)

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | The change after 2 weeks of intervention
  To measure pain intensity, The patients rated their pain level on an 11-point scale ranging from 0 to 10, which 0 indicates no pain and the highest score 10 indicates the worst possible pain

OTHER OUTCOMES:
The Oswestry disability index (ODI) | The change after 2 weeks of intervention
  This scale is self-assess questionnaire, which is designed to assess level of function and (disability) in activities of daily living in individual with LBP.It consists of ten everyday activities .A total score is calculated, percentage of disability (score obtained divided by 50 and multiplied by 100)
The Back Belief Questionnaire (BBQ) | The change after 2 weeks of intervention
  This is a specific self-report questionnaire consists of 14 items beliefs score help to Measuring back beliefs are associated with pain chronicity and disability in people with LBP.Score Range from 9 to 45 the higher the patients scores mean, the less he\she displays fear and false beliefs
physical performance test . | The change after 2 weeks of intervention
  six-minutes walking test , Repeated times sit to stand ,Repeated trunk flexion
Adherence to home exercise program | The patient commits to the intervention within 2 weeks
  diary to record every time they exercised

CONTACTS AND LOCATIONS:
Overall Officials: kholoud A Almufaireej, master, Principal Investigator — King saud unviersity
Locations (1):
- Security Forces Hospital, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Awaji, M. A. (2016). Epidemiology of low back pain in Saudi Arabia. Journal of Advances in Medical and Pharmaceutical Sciences, 1-9.
- [Background] Elbur, A. I. (2015). Level of adherence to lifestyle changes and medications among male hypertensive patients in two hospitals in Taif; Kingdom of Saudi Arabia. Int J Pharm Pharm Sci, 7(4), 168-172.
- [Result] Buchbinder R, van Tulder M, Oberg B, Costa LM, Woolf A, Schoene M, Croft P; Lancet Low Back Pain Series Working Group. Low back pain: a call for action. Lancet. 2018 Jun 9;391(10137):2384-2388. doi: 10.1016/S0140-6736(18)30488-4. Epub 2018 Mar 21. PMID 29573871
- [Result] Alamam DM, Moloney N, Leaver A, Alsobayel HI, Mackey MG. Pain Intensity and Fear Avoidance Explain Disability Related to Chronic Low Back Pain in a Saudi Arabian Population. Spine (Phila Pa 1976). 2019 Aug 1;44(15):E889-E898. doi: 10.1097/BRS.0000000000003002. PMID 30817741
- [Result] Leeuw M, Goossens ME, Linton SJ, Crombez G, Boersma K, Vlaeyen JW. The fear-avoidance model of musculoskeletal pain: current state of scientific evidence. J Behav Med. 2007 Feb;30(1):77-94. doi: 10.1007/s10865-006-9085-0. Epub 2006 Dec 20. PMID 17180640
- [Result] Garrett B, Taverner T, Masinde W, Gromala D, Shaw C, Negraeff M. A rapid evidence assessment of immersive virtual reality as an adjunct therapy in acute pain management in clinical practice. Clin J Pain. 2014 Dec;30(12):1089-98. doi: 10.1097/AJP.0000000000000064. PMID 24535053